CLINICAL TRIAL: NCT05752747
Title: The Effect of Shotblocker and Cold Massage on Pain, Crying Time and Physiological Parameters During Vaccine Injection in Babies
Brief Title: The Effect of Shotblocker and Cold Massage on Pain, Crying Time and Physiological Parameters in Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilek Kucuk Alemdar, Associate professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK 07
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Vaccine; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study was planned as randomized controlled experimental.
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to prevent selection bias, the assignment of infants to groups will be made using "stratification and randomization methods with blocks". Parents will not be informed which group their baby is in (ShotBlocker©, cold massage, control). In the study, the pain level of the infants will be evaluated by the family health worker, the researcher and their parents who administered the vaccine. At the end of the study, inter-observer agreement will be evaluated. Parents and family health workers will be informed by the researcher about the pain scale to be used in the research. In addition, the database of the research will be created by a university graduate statistician working in a statistical center independent of the research, apart from the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold Massage Group (Experimental): Just before the application, it will be taken out of the cabinet and the area to be vaccinated will be massaged with rollers with back and forth movements.
  Interventions: Other: Cold Massage Group
- ShotBlocker© Group (Experimental): It is a small flexible drug-free plastic tool. It is a small, flat-shaped instrument with a short, blunt, skin-contact ridge on the bottom and a hole in the center to inject. It is placed on the skin before injection. The protrusions on the inside do not harm the skin.
  Interventions: Other: ShotBlocker© Group
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Cold Massage Group — Just before the application, it will be taken out of the cabinet and the area to be vaccinated will be massaged with rollers with back and forth movements.
  Arms: Cold Massage Group
Other: ShotBlocker© Group — It is a small flexible drug-free plastic tool. It is a small, flat-shaped instrument with a short, blunt, skin-contact ridge on the bottom and a hole in the center to inject. It is placed on the skin before injection. The protrusions on the inside do not harm the skin.
  Arms: ShotBlocker© Group

SUMMARY:
The aim of this study is to determine the effect of ShotBlocker© and cold massage on pain, crying time and physiological parameters during DaBT-IPA-Hib vaccine administration in 2-6 months old babies.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of ShotBlocker© and cold massage on pain, crying time and physiological parameters during DaBT-IPA-Hib vaccine administration in 2-6 months old babies.This study was planned as randomized controlled experimental single-blind.

The population of the research will be 2-6 months old babies who come to Giresun Güce District State Hospital Family Health Center to receive DaBT-IPA-Hib vaccine between the dates of the research. The sample of the study will consist of infants who met the case selection criteria, accepted to participate in the study and were vaccinated between the specified dates.

As a result of the power analysis, it was determined that a total of 99 infants, 33 of whom were to be applied cold massage, 33 to be administered ShotBlocker©, and 33 to the control group, who were 2-6 months old to be administered DaBT-IPA-Hib vaccine, met the case selection criteria and agreed to participate in the study. Considering the possibility of case losses, a total of 108 babies, 36 in each group, are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* The baby is 2-6 months old,
* DaBT- IPA- Hib vaccine will be administered,
* The baby does not have a chronic disease,
* Parents must be at least primary school graduate,
* Parent's willingness to participate in the study.

Exclusion Criteria:

* Having a congenital or neurological health problem,
* Have taken an analgesic drug in the last 4 hours,
* Babies with a body temperature above 37.5 will not be included in the study.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
crying | 1 minute before the procedure
  crying time
crying | 1 minute after the procedure
  crying time will be measured and noted.
SpO2 | 1 minute before the procedure
  Physiological parameters
SpO2 | 1 minute after the procedure
  Physiological parameters
Pulse | 1 minute before the procedure
  Physiological parameters
Pulse | 1 minute after the procedure
  Physiological parameters
Body temperature | 1 minute before the procedure
  Physiological parameters
Body temperature | 1 minute after the procedure
  Physiological parameters
FLACC Pain Scale (Face, Legs, Activity, Cry, Consolability Pain Scale) | 1 minute before the procedure
  The FLACC scale was first developed by Merkel et al.in 1997. In the research, it will be used to evaluate the pain levels of infants in the experimental and control groups before, during and after vaccination. The five behaviors ("face", "legs", "activity", "crying" and "consolation") evaluated on this scale are considered indicators of pain that can be detected and graded by an observer. Descriptors for each item are accepted as indicators of children's painful behavior. Each item is scored from 0 to two, resulting in a pain intensity score ranging from 0 to 10. And descriptors associated with each score level represent pain intensity.
FLACC Pain Scale (Face, Legs, Activity, Cry, Consolability Pain Scale) | 1 minute after the procedure
  The FLACC scale was first developed by Merkel et al.in 1997. In the research, it will be used to evaluate the pain levels of infants in the experimental and control groups before, during and after vaccination. The five behaviors ("face", "legs", "activity", "crying" and "consolation") evaluated on this scale are considered indicators of pain that can be detected and graded by an observer. Descriptors for each item are accepted as indicators of children's painful behavior. Each item is scored from 0 to two, resulting in a pain intensity score ranging from 0 to 10. And descriptors associated with each score level represent pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Küçük Alemdar, Principal Investigator — Assoc. Dr.
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No